CLINICAL TRIAL: NCT06400927
Title: Safety of AI-Powered Virtual Assistant in Outpatient Management of Heart Failure: A Randomized Controlled Pilot Study: ASSIST-HF SIRIO
Brief Title: Safety of AI-Powered Virtual Assistant in Outpatient Management of Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: Clinical and Interventional Cardiology, Sassari University Hospital, Sassari, Italy (Unknown)
Responsible Party: Principal Investigator, Prof Diana Gorog, Professor, East and North Hertfordshire NHS Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RD2024-10
Record Dates: First submitted 2024-04-29; First posted 2024-05-06 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA-guided arm (Experimental)
  Interventions: Other: HF-guided VA
- Standard-of-care arm (Placebo Comparator)
  Interventions: Other: Standard-of-care

INTERVENTIONS:
Other: HF-guided VA — VA guided recommendation
  Arms: VA-guided arm
Other: Standard-of-care — Standard-of-care
  Arms: Standard-of-care arm

SUMMARY:
The aim of this pilot randomized study is to examine whether integrating the SIRIO-HF virtual assistant (VA) into the outpatient management of participants recently discharged from hospital with a new diagnosis of heart failure (HF), may reduce the need for regular medical assessment and the healthcare burden, reduce variability in healthcare, and meet with participant satisfaction, without compromising participant safety and overall care quality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Newly diagnosed HF with New York Heart Association class II-III symptoms at discharge

Exclusion Criteria

* Known prior history of HF
* Severe comorbidities that could affect protocol adherence, in the opinion of the investigator
* Alternative diagnosis for symptoms such as chronic obstructive pulmonary disease
* Dementia or other cognitive impairment
* Currently involved in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-06-13 (Estimated); Study Completion 2027-09-13 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the intervention to users (participants) | 12 weeks
  This will be assessed utilising an adapted 'acceptability of intervention measure' (AIM)

CONTACTS AND LOCATIONS:
Overall Officials: Diana A Gorog, MD, PhD, Principal Investigator — East and North Hertfordshire NHS Trust
Locations (1):
- East and North Hertfordshire NHS Trust, Stevenage, Hertfordshire, United Kingdom